CLINICAL TRIAL: NCT06110728
Title: Augmentation of Standard Psychotherapy With a Habit Change App: A Randomized Controlled Trial
Brief Title: Augmentation of Standard Psychotherapy With a Habit Change App
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of participant enrollment, the study was ended prematurely.
Sponsor: Rebecca Tavernier (Other)
Responsible Party: Sponsor-Investigator, Rebecca Tavernier, Senior Research Scientist, Weitzman Institute
Organization: Weitzman Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Habit change app
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetes; Substance Use Disorders; Anxiety Disorders; Depression
Keywords: mobile health; randomized control trial; mental health; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Substance-Related Disorders; Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants with a diagnosis of diabetes and depression, anxiety, and/or substance use disorder will be randomized to one of two treatment groups: (1) Habit Change and (2) TAU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habit Change (Experimental): Participants randomly assigned to the Habit Change arm will be asked to track behaviors related to their specific goals on a daily basis through the app and will be allowed to engage with the app freely. Outside of using the app, participants will not be asked to engage in any additional activities beyond those typically engaged in for behavioral health treatment (e.g., completion of mental and behavioral health outcome measures).
  Interventions: Behavioral: Habit Change
- Treatment as Usual (No Intervention): Participants in the TAU arm will continue to engage in their behavioral health treatment as usual and will not be provided access to the habit change app.

INTERVENTIONS:
Behavioral: Habit Change — Participants assigned to the Habit Change arm will be asked to track behaviors related to their specific goals on a daily basis through the app and will be allowed to engage with the app freely. Goals can include things like reaching a step goal, sleeping for a certain number of hours, or making healthy food choices.
  Arms: Habit Change

SUMMARY:
The goal of this clinical trial is to document the efficacy of using a habit change application (app) as an adjunct to standard psychotherapy among individuals with diabetes receiving mental health treatment for depression, anxiety, or substance use disorders. The main questions it aims to answer are:

Question 1: When behavioral health treatment is augmented with a habit change app for between visit care, does the use of this tool improve mental and behavioral health outcomes?

Question 2: Are there certain populations who benefit more from using a habit change app?

Question 3: Does use of a habit change app impact healthcare utilization and costs?

Exploratory Research Question: Does use of a habit change app impact physical health outcomes, including A1c levels, blood pressure, and weight?

Participants selected to receive the habit change app will be asked to track goals that they set for themselves in adjunct to their current behavioral health treatment; those selected for treatment as usual will have no additional steps to take. Researchers will compare the groups to see if there are different outcomes in symptom reports and healthcare utilization.

DETAILED DESCRIPTION:
As part of this research, participants with a diagnosis of diabetes and depression, anxiety, and/or substance use disorder will be randomized to one of two treatment groups: (1) Habit Change and (2) Treatment as Usual (TAU). All participants will currently be engaged in behavioral health treatment. Participants in the Habit Change arm will obtain access to a habit change app and set their personal health goals in the app to track throughout the study period. Participants in the TAU arm will continue to engage in their behavioral health treatment as usual and will not be provided access to the habit change app. Participants randomly assigned to the Habit Change arm will be asked to track behaviors related to their specific goals on a daily basis through the app and will be allowed to engage with the app freely. Outside of using the app, participants will not be asked to engage in any additional activities beyond those typically engaged in for behavioral health treatment (e.g., completion of mental and behavioral health outcome measures).We will be recruiting up to 600 participants as part of this research study (300 per treatment arm).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 Diabetes
* Are being seen by a clinician for depression, anxiety and/or substance use disorder
* Speak English
* Have an Apple device to download the habit change app

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Changes in depression ratings | Enrollment and up to 3 months following enrollment
  Participants will report their depressive symptoms using the Patient Health Questionnaire-9 (PHQ-9) prior to each individual therapy session. Changes in depression scores from baseline to the end of the study period (up to 3 months after enrollment) will be evaluated. The PHQ-9 is a validated self-report measure assessing depressive symptoms over the previous 2 weeks. The PHQ-9 total score ranges from 0 to 27, with higher scores indicating worse depressive symptoms (scores of 0-4 are classified as minimal depression; 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; and ≥ 20 as severe depression).
Changes in anxiety ratings | Enrollment and up to 3 months following enrollment
  Participants will report their anxiety symptoms using the Generalized Anxiety Disorder-7 (GAD-7) measure prior to each individual therapy session. Changes in anxiety scores from baseline to the end of the study period (up to 3 months after enrollment) will be evaluated. The GAD-7 is a validated self-report measure assessing anxiety symptoms over the previous 2 weeks. The GAD-7 total score ranges from 0 to 21, with higher scores indicating worse anxiety symptoms (scores of 0-4 are classified as minimal anxiety; 5-9 are classified as mild anxiety; 10-14 as moderate anxiety; and ≥ 15 as severe anxiety).
Number of billable visits attended | Enrollment through up to three months following enrollment
  Healthcare utilization (i.e., number of billable visits attended) will be extracted from the electronic health record for each participant at the end of the study period. The number of billable visits participants attended over the course of the study period (up to 3 months) will be compared between treatment groups.
Number of missed behavioral health visits | Enrollment through up to three months following enrollment
  The number of missed behavioral health visits will be extracted from the electronic health record for each participant at the end of the study period. The number of missed behavioral health visits over the course of the study period (up to 3 months) will be compared between treatment groups.

OTHER OUTCOMES:
Changes in A1c levels | Enrollment and up to 3 months following enrollment
  A1c readings will be extracted from the electronic health record at the time of enrollment and the end of the study period (up to three months after enrollment) for each participant. Changes in A1c level from enrollment to the end of the study period will be compared between treatment groups.
Changes in blood pressure | Enrollment and up to 3 months following enrollment
  Blood pressure readings will be extracted from the electronic health record at the time of enrollment and the end of the study period (up to three months after enrollment) for each participant. Changes in blood pressure from enrollment to the end of the study period will be compared between treatment groups.
Changes in weight | Enrollment and up to 3 months following enrollment
  Measured weight (in kilograms) will be extracted from the electronic health record at the time of enrollment and the end of the study period (up to three months after enrollment) for each participant. Changes in weight from enrollment to the end of the study period will be compared between treatment groups.

IPD SHARING:
Plan to Share IPD: No